CLINICAL TRIAL: NCT04209478
Title: Transversus Abdominis Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia in Pediatric Patients; a Prospective, Randomized, Controlled Study
Brief Title: Transversus Abdominis Plane Block and Quadratus Lumborum Block in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BakirkoySadiKonu
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative
Keywords: quadratus lumborum block; pediatric anesthesia; transverse abdominal block
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block (Experimental): Cases were assessed transversus abdominis plane block for postoperative analgesia
  Interventions: Drug: Tramadol hydrochloride
- QL Block (Experimental): Cases were assessed quadratus lumborum block for postoperative analgesia
  Interventions: Drug: Tramadol hydrochloride

INTERVENTIONS:
Drug: Tramadol hydrochloride — The Wong-Baker facial pain scale was used to assess pain (1: no pain, 10: worst possible pain). During monitoring patients with pain score ≥3 had intravenous 1 mg/kg tramadol hydrochloride administered, After 15 minutes following tramadol injection, cases with pain score continuing ≥3 were to be assessed as insufficient analgesia and had 0.1 mg/kg morphine hydrochloride planned for intravenous administration
  Other Names: morphine hydrochloride

SUMMARY:
In the pediatric age group, postoperative pain is very important for the children to have a comfortable and problem-free postoperative period.

In the present study, it was aimed to compare the postoperative analgesic efficacy of Transversus abdominis plane (TAP) Block, and quadratus lumborum block (QLB) Type 1 on the pediatric patients

DETAILED DESCRIPTION:
Patients included in the study were randomly divided into 2 groups. Cases were assessed ultrasonography-guided TAP block (Group B, n=20) or ultrasonography-guided QL Block. Total analgesic amounts in 24 hours and first analgesic requirement times recorded.

ELIGIBILITY:
Inclusion Criteria:

* The study included 40 cases undergoing lower abdominal surgery aged from 3 to 16 years with American Society of Anesthesiologist I-II level.

Exclusion Criteria:

* Cases with American Society of Anesthesiologist III-IV health level and those with a history of allergy to local anesthetic medications were not included in the study

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-30 (Actual); Study Completion 2016-11-30 (Actual)

PRIMARY OUTCOMES:
the analgesic use of the groups in 24 hours | how many times in 24 hours
  the number of analgesic requirements

CONTACTS AND LOCATIONS:
Locations (1):
- Döndü Genç Moralar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Blanco+R%2C+Ansari+T%2C+Riad+W%2C+Shetty+N.+Quadratus+Lumborum+Block+Versus+Transversus+Abdominis+Plane+Block+for+Postoperative+Pain+After+Cesarean+Delivery.